CLINICAL TRIAL: NCT01199562
Title: Modified Preemptive CMV Management Strategy After Allogeneic Hematopoietic Cell Transplantation and Laboratory Correlation With Innate Immune Function
Brief Title: Infection Prophylaxis and Management in Treating Cytomegalovirus (CMV) Infection in Patients With Hematologic Malignancies Previously Treated With Donor Stem Cell Transplant
Status: Active, not recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 09038; NCI-2010-01932
Record Dates: First submitted 2010-09-08; First posted 2010-09-13 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic/Lymphoid Cancer; Accelerated Phase Chronic Myelogenous Leukemia; Acute Undifferentiated Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Grade III Lymphomatoid Granulomatosis; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Aplastic Anemia; Atypical Chronic Myeloid Leukemia, BCR-ABL Negative; Blastic Phase Chronic Myelogenous Leukemia; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; Contiguous Stage II Adult Burkitt Lymphoma; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Contiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Contiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Contiguous Stage II Adult Lymphoblastic Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Cytomegalovirus Infection; de Novo Myelodysplastic Syndromes; Essential Thrombocythemia; Extramedullary Plasmacytoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Isolated Plasmacytoma of Bone; Mast Cell Leukemia; Meningeal Chronic Myelogenous Leukemia; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Polycythemia Vera; Post-transplant Lymphoproliferative Disorder; Previously Treated Myelodysplastic Syndromes; Primary Myelofibrosis; Primary Systemic Amyloidosis; Progressive Hairy Cell Leukemia, Initial Treatment; Prolymphocytic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Secondary Myelofibrosis; Splenic Marginal Zone Lymphoma; Stage 0 Chronic Lymphocytic Leukemia; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Mixed Cell Lymphoma; Stage I Adult Diffuse Small Cleaved Cell Lymphoma; Stage I Adult Hodgkin Lymphoma; Stage I Adult Immunoblastic Large Cell Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Adult T-cell Leukemia/Lymphoma; Stage I Chronic Lymphocytic Leukemia; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Multiple Myeloma; Stage I Mycosis Fungoides/Sezary Syndrome; Stage I Small Lymphocytic Lymphoma; Stage II Adult Hodgkin Lymphoma; Stage II Adult T-cell Leukemia/Lymphoma; Stage II Chronic Lymphocytic Leukemia; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma; Stage II Multiple Myeloma; Stage II Mycosis Fungoides/Sezary Syndrome; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; T-cell Large Granular Lymphocyte Leukemia; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Anemia, Aplastic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Cytomegalovirus Infections; Thrombocythemia, Essential; Intraocular Lymphoma; Leukemia, Mast-Cell; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Polycythemia Vera; Primary Myelofibrosis; Immunoglobulin Light-chain Amyloidosis; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — Therapeutics; Flow Cytometry; Ganciclovir; Valganciclovir; Foscarnet; Antiviral Agents; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Arm I: Patients receive standard antiviral infection prophylaxis and management comprising ganciclovir, valganciclovir, or foscarnet sodium for 2 weeks or until the plasma CMV DNA Q-PCR is negative. Patients may receive additional courses based on subsequent CMV reactivations.
  Interventions: Procedure: infection prophylaxis and management; Other: laboratory biomarker analysis; Other: flow cytometry; Genetic: DNA analysis; Genetic: RNA analysis; Procedure: management of therapy complications; Drug: ganciclovir; Drug: valganciclovir; Drug: foscarnet sodium; Procedure: antiviral therapy; Genetic: polymerase chain reaction; Genetic: protein expression analysis

INTERVENTIONS:
Procedure: infection prophylaxis and management — Undergo infection prophylaxis and management
  Other Names: treatment of infectious disease
Other: laboratory biomarker analysis — Correlative studies
Other: flow cytometry — Correlative studies
Genetic: DNA analysis — Correlative studies
Genetic: RNA analysis — Correlative studies
Procedure: management of therapy complications — undergo infection prophylaxis and management
  Other Names: complications of therapy, management of
Drug: ganciclovir — Given IV
  Other Names: BW 759U; BW-B759U
Drug: valganciclovir — Given orally
  Other Names: Valcyte; VGCV
Drug: foscarnet sodium — Given orally
  Other Names: Foscavir; trisodium phosphonoformate
Procedure: antiviral therapy — undergo infection prophylaxis and management
  Other Names: therapy, antiviral
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
Genetic: protein expression analysis — Correlative studies

SUMMARY:
RATIONALE: Infection prophylaxis and management may help prevent cytomegalovirus (CMV) infection caused by a stem cell transplant.

PURPOSE:This clinical trial studies infection prophylaxis and management in treating cytomegalovirus infection in patients with hematologic malignancies previously treated with donor stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy and safety of a individualized strategy for cytomegalovirus (CMV) preemptive management, one that monitors CMV viral load and clinical markers of immunosuppression to optimize use of ganciclovir in recipients of allogeneic hematopoietic cell transplantation (HCT) who experience CMV reactivation.

SECONDARY OBJECTIVES:

I. To investigate how donor killer-cell immunoglobulin-like receptors (KIR) genes of interest (activating KIR2DS2 and 2DS4, inhibitory KIR2DL1, 2DL2/2DL3, 3DL1, 3DL2), together with their recipient ligands where known, influence CMV reactivation-free survival after allogeneic HCT, independently of clinical risk factors such as onset of acute graft-versus-host disease.

II. To investigate whether markers of natural killer (NK) cell function correlate with a) KIR/ligand compound genotype and baseline or concurrent clinical factors and b) with history of CMV reactivation and anti-CMV therapy at the time of NK cell collection.

III. To investigate associations between NK cell recovery and antigen-specific T cell immune reconstruction.

OUTLINE: Patients receive standard antiviral infection prophylaxis and management comprising ganciclovir, valganciclovir, or foscarnet sodium for 2 weeks or until the plasma CMV deoxyribonucleic acid (DNA) quantitative polymerase chain reaction (Q-PCR) is negative. Patients may receive additional courses based on subsequent CMV reactivations.

After completion of study treatment, patients are followed up for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: hematologic malignancies/disorders including aplastic anemia and myelodysplastic syndrome
* Procedure: first allogeneic, T cell-replete transplantation of stem-cells from peripheral blood or bone marrow of an human leukocyte antigen (HLA) matched, unrelated or nonsyngeneic sibling donor
* CMV seropositive donor and/or recipient
* Performance level: must have already been determined to be eligible for HCT at City of Hope (COH)
* Organ function requirements: The minimum organ function requirements should be the same as the requirements for HCT
* Informed Consent: All patients must be capable of signing a written informed consent and no consent can be provided by a legal guardian

Exclusion Criteria:

* The recipient had prior polymerase chain reaction (PCR) positive CMV infection in blood or organ-specific disease in the past 12 months
* The source of hematopoietic stem cells is T-cell depleted
* Concomitant anti-graft-versus-host disease (GVD) treatment includes in vivo T cell depletion
* Recipient is human immunodeficiency virus (HIV)-1 positive
* No prior allogeneic HCT (Allo HCT) (autologous HCT [Auto HCT] is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12-30 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Initiation of anti-CMV therapy | Day 80 post stem cell transplant
  Subjects will not be considered treated with anti-CMV agents unless at least 4 consecutive days of therapy are completed.
Diagnosis of CMV pneumonia | 1 year
  Confirmed by detection of CMV in bronchoalveolar lavage or lung biopsy. Reported overall and separately for those whose preemptive management was and was not modified (postponed or foregone or limited to a false start) and compared to corresponding incidence in a similar cohort at our institution.

SECONDARY OUTCOMES:
CMV reactivation-free survival, monitored using a real time PCR assay for CMV DNA in plasma | Up to day 100 post-transplant
  Modeled using proportional hazards regression. Primary risk factors will be donor KIR of interest (activating KIR2DS2 and 2DS4, inhibitory KIR2DL1, 2DL2/2DL3, 3DL1, 3DL2), together with their recipient ligands where known. Potential confounding factors to be controlled in the model will include established clinical risk factors, including pretransplant CMV serostatus of donor and recipient, unrelated donor, marrow versus peripheral blood stem cells, and onset of acute graft-versus-host disease, handled as a time-dependent variable. The proportionality of hazards over time will be verified.
Percent cytotoxicity and ex vivo percent CD56+/CD107B+ cells | Day 120 post stem cell transplant
  Studied longitudinally in generalized linear models. Each of the 2 markers of NK function will be modeled separately.

CONTACTS AND LOCATIONS:
Overall Officials: Ryotaro Nakamura, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States